CLINICAL TRIAL: NCT04813380
Title: Serum MicroRNAs 223 and 146a in Allergic Rhinitis Patients: Correlation With Disease Severity and Their Role as Biomarkers for Efficacy of Sublingual Immunotherapy
Brief Title: Serum MicroRNAs 223 and 146a in Allergic Rhinitis Patients as Biomarkers for Efficacy of Sublingual Immunotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Fatma Zohry Kamel Khater, Dr, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Sublingual immunotherapy
Record Dates: First submitted 2021-03-20; First posted 2021-03-24 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Effects of Immunotherapy
Keywords: Allergen immunotherapy; MiRNA-223; MiRNA-146a
MeSH Terms: interventions — Sublingual Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oraltek Sublingual immunotherapy group (Active Comparator): one drops under tongue for ten days then three Drops for another ten days then five drops for another ten days for three successive months then five drops every two days per week for two months then five drops one day per week for one months
  Interventions: Other: Sublingual immunotherapy
- Placebo (Placebo Comparator): one drops under the tongue then three drops then five drops for three successive months then five drops every two days per week for two months then five drops one day per week for one months
  Interventions: Other: Sublingual immunotherapy

INTERVENTIONS:
Other: Sublingual immunotherapy — Sublingual immunotherapy give to allergic rhinitis patients for treatment

SUMMARY:
The aim of the study is:

* to evaluate the serum levels of miR-223 and miRNA146a and to assess their correlation with disease severity in allergic rhinitis patients and their role as biomarkers for efficacy of sublingual immunotherapy.
* also to find if high sensitivity CRP can be an easy non-expensive test for diagnosis and follow up of allergic rhinitis patients.

DETAILED DESCRIPTION:
Over the last decades the prevalence of allergic disease has steadily been rising and recent figures indicate that in the western world 10-25% of people are affected with allergic diseases ranging from food allergy, atopic dermatitis/ eczema, allergic rhinitis, hay fever to asthma.

Allergic rhinitis (AR) is the most frequent allergic disease in Western Europe that interferes with school attendance and performance, with a prevalence rate of 20-30%. Very few studies of the epidemiology were done about the prevalence of allergic rhinitis in Egypt as its prevalence was 9 %.

Allergic rhinitis is allergen-specific IgE-mediated inflammatory reactions which is characterized by excessive eosinophil infiltration, Th2 cytokine responses such as IL5, IL4, IL13, and mucus secretion. The prevalence of allergic rhinitis is increasing worldwide due to changes in the socioeconomic status, environmental factor, and occupational factor. AR burden on sleep and learning is substantial in children. Moreover, AR is considered a risk factor for subsequent asthma comorbidity.

Allergic rhinitis is characterized by nasal congestion, itching, rhinorrhea, and sneezing, which are manifested as a consequence of inappropriate immune responses mediated by allergen specific immunoglobulin E (IgE) antibodies toward otherwise harmless antigens such as pollen and house dust mite (HDM).

High-sensitivity-C-reactive protein (hs-CRP) is a well-known systemic inflammatory marker that is easy and inexpensive to measure, together with ESR, serum Ig-E and total eosinophil count are measured as laboratory markers of allergic diseases.

MicroRNAs (miRNAs) are small non-coding RNA molecules that are 18-22 nucleotides long and highly conserved throughout evolution. MiRNAs play important roles in numerous disease processes such as asthma and allergic rhinitis and that differential miRNA expression can identify novel subtypes of these diseases. As approximately 150 miRNAs are detectable in the blood, differential miRNA expression patterns may serve as a molecular fingerprint that aids in disease diagnosis, characterization, and prognosis.

MiRNAs may have particular clinical utility in allergic diseases. These diseases are characterized by tissue inflammation and are particularly difficult to diagnose and characterize considering that measuring releasing mediators, such as cytokines in blood which their characteristic measurement is unreliable . As a result, invasive methods (e.g., bronchoscopy and tissue biopsies) are needed to quantify inflammatory changes. It follows that miRNA expression profiling in blood and other body fluids becomes important for identifying and developing novel, non-invasive disease Biomarkers.

One of the most significantly upregulated molecules was miR-223 involved in eosinophilic inflammation and associated with lower regulatory T-cell numbers. It is well known that Treg cells play an important role in development of tolerance by producing IL-10. Thus, in the future inhibition of miR-223 could be considered an adjuvant treatment.

MiR-146a is one of the two members of the miR-146 miR family. It has been reported to be involved in a large number of cell activi¬ties, such as suppression of cancer growth, inhibition of inflam¬mation, regulation of the immune system and suppression of allergic inflammation. MiR-146a play a role in regulation of allergic diseases such as allergic rhinitis by modulating Treg cells.

Allergen-specific immunotherapy (AIT) is currently the only known causal effective treatment of IgE-mediated allergy. Sublingual immunotherapy is a well-established allergen-specific immunotherapy and a safe and effective strategy to reorient inappropriate immune responses in allergic patients.

MiR-146a may play a role in allergen immunotherapy of allergic diseases by modulating Treg cells. Also., high miR-223 expression is associated with lower regulatory T-cell numbers.

ELIGIBILITY:
Inclusion Criteria:

1. Patient consent.
2. Patients between 6-60 years old suffering from allergic rhinitis clinically.
3. Positive skin prick test

Exclusion Criteria:

* 1- Chronic inflammatory condition as COPD, tuberculosis, aspergillosis and chronic hepatitis.

  2- Other allergic diseases as bronchial asthma, allergic conjunctivitis and chronic urticaria 3- Those undergoing chronic treatment with systemic steroids or B- blockers 4- Systemic immunological disorders as systemic lupus erythematous, rheumatoid arthritis and systemic sclerosis.

  5- Malignancy

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
MiRNA146a, microRNA 223 measurements | 6 months
  Effect of sublingual immunotherapy on the miRNA146, MicroRNA 223 on allergic rhinitis patients

CONTACTS AND LOCATIONS:
Locations (1):
- Fatma Zohry Kamel Khater, Zagazig, Egypt

REFERENCES:
- [Background] Joint Task Force on Practice Parameters; American Academy of Allergy, Asthma and Immunology; American College of Allergy, Asthma and Immunology; Joint Council of Allergy, Asthma and Immunology. Allergen immunotherapy: a practice parameter second update. J Allergy Clin Immunol. 2007 Sep;120(3 Suppl):S25-85. doi: 10.1016/j.jaci.2007.06.019. No abstract available. PMID 17765078
- [Background] Gebert LFR, MacRae IJ. Regulation of microRNA function in animals. Nat Rev Mol Cell Biol. 2019 Jan;20(1):21-37. doi: 10.1038/s41580-018-0045-7. PMID 30108335
- [Background] Hosseini SA, Zilaee M, Shoushtari MH, Ghasemi Dehcheshmeh M. An evaluation of the effect of saffron supplementation on the antibody titer to heat-shock protein (HSP) 70, hsCRP and spirometry test in patients with mild and moderate persistent allergic asthma: A triple-blind, randomized placebo-controlled trial. Respir Med. 2018 Dec;145:28-34. doi: 10.1016/j.rmed.2018.10.016. Epub 2018 Oct 19. PMID 30509713
- [Background] Hou B, Murata M, Said AS, Sakaida H, Masuda S, Takahashi T, Zhang Z, Takeuchi K. Changes of micro-RNAs in asymptomatic subjects sensitized to Japanese cedar pollen after prophylactic sublingual immunotherapy. Allergy Rhinol (Providence). 2015 Jan;6(1):33-8. doi: 10.2500/ar.2015.6.0107. Epub 2015 Feb 11. PMID 25675113
- [Background] Jay DC, Nadeau KC. Immune mechanisms of sublingual immunotherapy. Curr Allergy Asthma Rep. 2014 Nov;14(11):473. doi: 10.1007/s11882-014-0473-1. PMID 25195100
- [Background] Jutel M, Kosowska A, Smolinska S. Allergen Immunotherapy: Past, Present, and Future. Allergy Asthma Immunol Res. 2016 May;8(3):191-7. doi: 10.4168/aair.2016.8.3.191. PMID 26922928
- [Background] Levy BD, Kohli P, Gotlinger K, Haworth O, Hong S, Kazani S, Israel E, Haley KJ, Serhan CN. Protectin D1 is generated in asthma and dampens airway inflammation and hyperresponsiveness. J Immunol. 2007 Jan 1;178(1):496-502. doi: 10.4049/jimmunol.178.1.496. PMID 17182589
- [Background] Luo X, Hong H, Tang J, Wu X, Lin Z, Ma R, Fan Y, Xu G, Liu D, Li H. Increased Expression of miR-146a in Children With Allergic Rhinitis After Allergen-Specific Immunotherapy. Allergy Asthma Immunol Res. 2016 Mar;8(2):132-40. doi: 10.4168/aair.2016.8.2.132. Epub 2015 Oct 22. PMID 26739406
- [Background] Moustafa Y, El Nady HG, Saber MM, Dabbous OA, Kamel TB, Abel-Wahhab KG, Sallam SF, Zaki DA. Assessment of Allergic Rhinitis among Children after Low-Level Laser Therapy. Open Access Maced J Med Sci. 2019 Jun 30;7(12):1968-1973. doi: 10.3889/oamjms.2019.477. eCollection 2019 Jun 30. PMID 31406538
- [Background] Panganiban RP, Pinkerton MH, Maru SY, Jefferson SJ, Roff AN, Ishmael FT. Differential microRNA epression in asthma and the role of miR-1248 in regulation of IL-5. Am J Clin Exp Immunol. 2012 Nov 15;1(2):154-65. Print 2012. PMID 23885321
- [Background] Panganiban RP, Lambert KA, Hsu MH, Laryea Z, Ishmael FT. Isolation and profiling of plasma microRNAs: Biomarkers for asthma and allergic rhinitis. Methods. 2019 Jan 1;152:48-54. doi: 10.1016/j.ymeth.2018.06.007. Epub 2018 Jun 12. PMID 29906503
- [Background] Platts-Mills TA. The allergy epidemics: 1870-2010. J Allergy Clin Immunol. 2015 Jul;136(1):3-13. doi: 10.1016/j.jaci.2015.03.048. PMID 26145982
- [Background] Specjalski K, Jassem E. MicroRNAs: Potential Biomarkers and Targets of Therapy in Allergic Diseases? Arch Immunol Ther Exp (Warsz). 2019 Aug;67(4):213-223. doi: 10.1007/s00005-019-00547-4. Epub 2019 May 28. PMID 31139837
- [Background] Zhao Y, Zhao Y, Zhang Y, Zhang L. HLA-II genes are associated with outcomes of specific immunotherapy for allergic rhinitis. Int Forum Allergy Rhinol. 2019 Nov;9(11):1311-1317. doi: 10.1002/alr.22384. Epub 2019 Jul 12. PMID 31299142